CLINICAL TRIAL: NCT02786082
Title: Single Center, Randomized, Open Labeled Pharmacokinetics Study of Azilsartan Tablets in Chinese Healthy Volunteers
Brief Title: Pharmacokinetics Study of Azilsartan Tablets in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zhaoke-201603-Azil
Record Dates: First submitted 2016-05-24; First posted 2016-05-30 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — azilsartan

ARMS (2):
- Group I (Experimental): For Pharmacokinetics Studies of Azilsartan with Single-dose oral administration, 12 subjects in group I, half are male and half are female, will take Azilsartan tablet 20mg orally on fasting.
  For Pharmacokinetics Studies of Azilsartan with Multiple-dose oral administration, 12 subjects in group I will take 20mg Azilsartan orally once daily for 7 day (day 3~day 9) after completing the last time blood sample collection (in day 2, 48h) of the first time administration (day 1)
  Interventions: Drug: 20mg Azilsartan Tablets
- Group II (Experimental): For Pharmacokinetics Studies of Azilsartan with Single-dose oral administration, 12 subjects in group II, half are male and half are female, will take Azilsartan tablet 40mg orally on fasting.
  For The effects of diet for pharmacokinetic study: The 12 healthy subjects, in group II (in single-dose administration study), after 7-day washout period after the first administration (at day 1, 40mg) will receive Azilsartan tablet 40mg after high-fat diet at day 8
  Interventions: Drug: 40mg Azilsartan Tablets

INTERVENTIONS:
Drug: 20mg Azilsartan Tablets — Strength: 20mg, oral administration 1 tablet/ day
  Arms: Group I
Drug: 40mg Azilsartan Tablets — Strength: 40mg, oral administration 1 tablet/ day
  Arms: Group II

SUMMARY:
The main objective is to study the pharmacokinetics of Azilsartan Tablets in human and providing evidence for clinical study and clinical application of this product.

DETAILED DESCRIPTION:
This is a Single center, randomized, open labeled study. The study is conducted to evaluate the pharmacokinetics Studies of Azilsartan with single-dose oral administration, multiple-dose oral administration and effects of diet.

1) Pharmacokinetics Studies of Azilsartan with Single-dose oral administration: 24 healthy subjects will be randomly divided into 2 groups evenly, Group I and Group II, with 12 subjects in each group, half are male and half are female. Group I will take Azilsartan tablet 20mg orally on fasting, while Group II will take Azilsartan tablet 40mg orally on fasting. Blood sampling time: 0h (before administration starting), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48h after administration. 5ml whole blood from cubital vein will be placed in a heparinized tube and centrifuged. Duplicated plasma A and B will be taken and kept in low temperature.

2）Pharmacokinetic Studies of Azilsartan Tablets with Multiple-dose oral administration Subjects in Group I will take 20mg Azilsartan orally once daily for 7 day (day 3~day 9) after completing the last time blood sample collection (in day 2, 48h) of the first time administration (day 1). 5mL blood sample will be collected from vein on day 7, day 8 and day 9 for measuring minimum observed concentration before drug administration. On day 9, after administration, blood sampling time is the same as single-dose administration study. Blood sampling time: 0h (before administration starting), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48h after administration. 5ml whole blood from cubital vein will be placed in a heparinized tube and centrifuged. Duplicated plasma A and B will be taken and kept in low temperature.

3）The effects of diet for pharmacokinetic study: The 12 healthy subjects, in group II (in single-dose administration study), after 7-day washout period after the first administration (at day 1, 40mg) will receive Azilsartan tablet 40mg after high-fat diet at day 8, and the blood sampling time point after administration is the same as in single-dose administration study. The process, storage condition of the blood samples are the same as single-dose administration study. Blood sampling time: 0h (before administration starting), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48h after administration. 5ml whole blood from cubital vein will be placed in a heparinized tube and centrifuged. Duplicated plasma A and B will be taken and kept in low temperature.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects in all groups will be adult females or adult males between 18 and 45 (inclusive) years of age, the year age difference between each subject cannot be more than 10.
2. Body mass index (BMI) within the range 19~25kg/m2 (inclusive). BMI=weight (kg)/height(m)2。
3. Subjects are eligible to participate if the results of physical examination （height, weight, respiration, pulse, blood pressure, thorax, abdomen, etc） and laboratory examination (blood routine examination, urine routine test, blood chemistry test, infectious disease screening, etc) are normal, the tests above will be conducted to all the subjects before the trial initiating. The results of ECG and chest X-ray are normal or slightly abnormal without clinical significance.
4. Subjects should not have history of cardiovascular disease, liver disease, renal disease, digestive disease, psychiatric disease, neuropathy disease, etc.
5. Subjects who do not have allergic history of Angiotensin Receptor Blockers, the other drugs and biological agents.
6. Subjects who are not addicted to smoking and alcohol and without the other bad habits.
7. Subjects have not participated in other clinical trial and donated blood within 3 months prior to this trial,
8. Subjects have well known the nature, significance, possible benefits, inconveniences and potential risks before participating in this trial and understood the trial process. Subjects are voluntary to participate in this trial.

Exclusion Criteria:

1. Subjects who have abnormalities with clinical significance in physical examination, laboratory examination, 12-lead ECGs, chest X-ray.
2. Subjects with history of orthostatic hypotension, gastrointestinal disease (such as gastric ulcer, gastritis, etc), renal disease (such as nephritis, nephropyelitis, etc), or cardiovascular, respiratory, neurological, psychotic, haematological, endocrine or the other disorders.
3. Subjects with allergic constitution with history of sensitivity to Angiotensin Receptor Blockers or a history of the other drugs and biological agent.
4. Systolic blood pressure (SBP) <90mmHg or >140mmHg, and/or diastolic blood pressure (DBP) <50mmHg or >90mmHg. Subjects with orthostatic hypotension (at screening, symptomatic or asymptomatic orthostatic hypotension is defined as: subject lying down comfortably for 5 minutes, the blood pressure which is recorded at 5 min considered to be the baseline. The time point of subject stands is considered to be the onset time. Orthostatic hypotension is diagnosed by a rise in systolic blood pressure of 20mmHg or more, or a decrease in diastolic blood pressure of 20mmHg or more, when standing with arms relaxing).
5. Vegetarian.
6. Subjects who plan to bear children in 6 months.
7. History of alcohol abuse in the last 6 months prior to screening defined as an average weekly intake of greater than 14 unit (one unit is equivalent to 360ml of beer or 45ml of spirits with 40% alcohol content or 150 ml of wine). History of smoking >5 cigarettes a day in the last 6 months prior to screening.
8. History of administrating any drugs that will effect this trial. Subjects who have participated in donation of blood or any drug clinical trial(as subjects) in the last 3 months, or are taking any other drugs.
9. Hepatitis B patients, or Hepatitis C patients, or hepatitis C carrier, or subjects with immunodeficiency, or positive HIV antibody results, or positive syphilis antibody results.
10. 72 hours prior to randomization, subjects with history of special diet (includes grapefruit, xanthine diet, chocolate, caffeinated coffee or tea, or any other caffeinated beverages) or strenuous exercise, or with the other factors that will effect the absorption, distribution, metabolism and excretion.
11. Subjects who took prescription drugs 2 weeks before study.
12. Subjects who, in the opinion of the investigators, should not participate in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | Pre-dose, 15 minutes, 30 minutes, 1 hour, 1.5 hour , 2 hours, 2.5 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 16 hours, 24 hours, 36 hours, 48 hours after administration
  To observe area under curve characteristics of Azilsartan in 20mg and 40mg single dose and 20mg multiple dose groups
Area Under Curve (AUC) | Pre-dose, 15 minutes, 30 minutes, 1 hour, 1.5 hour , 2 hours, 2.5 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 16 hours, 24 hours, 36 hours, 48 hours after administration
  To observe area under curve characteristics of Azilsartan in fasting and high fat diet group